CLINICAL TRIAL: NCT01467440
Title: Efficacy of Selective Laser Trabeculoplasty in Patients Under Treatment With Topical Prostaglandines
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SLT_PG_2011
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma and Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- PGA: Patients under glaucoma treatment with prostaglandines
  Interventions: Device: Selective Laser Trabeculoplasty
- NON-PGA: Patient not recieving prostaglandines to treat their glaucoma
  Interventions: Device: Selective Laser Trabeculoplasty

INTERVENTIONS:
Device: Selective Laser Trabeculoplasty — trabeculoplasty with an SLT-Laser to reduce intraocular pressure
  Other Names: SLT-Laser, Tango Laser, Ellex Medical Pty. Ltd., 82 Gilbert Street, Adelaide, SA 5000 Australia

SUMMARY:
Retrospective analysis of efficacy of selective laser trabeculoplasty in patients under treatment with topical prostaglandins compared to patients without topical prostaglandins is performed.

Inclusion criterion are patients with glaucoma or ocular hypertension, who underwent treatment with selective laser trabeculoplasty due to insufficient control of intraocular pressure during their routine treatment at the University Hospital Zurich / Division of Ophthalmology.

ELIGIBILITY:
Inclusion criteria:

* Patients with ocular hypertension or glaucoma who underwent selective laser trabeculoplasty due to insufficient control of intraocular pressure despite maximum tolerated topical treatment.

Exclusion criteria:

* Optic neuropathy other than glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
IOP | t0

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Jens Funk, Professor, MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland